CLINICAL TRIAL: NCT07204483
Title: Community-Based Feasibility Trial Comparing Functional Clothing, Moderate Exercise, and Health Information for Stress Reduction and Behavior Change in Adults in Yomitan Village, Okinawa, Japan
Brief Title: Feasibility Trial of Functional Clothing, Moderate Exercise, and Health Information for Stress Reduction and Behavior Change in Okinawa
Acronym: Y-RELIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shinyu Kise (Other)
Responsible Party: Sponsor-Investigator, Shinyu Kise, Director, Institute for Tourism and Health; Principal Investigator, Ryusei Hospital, General Incorporated Foundation Ryukyuseimeisaiseikai, Ryusei Hospital.
Organization: General Incorporated Foundation Ryukyuseimeisaiseikai, Ryusei Hospital. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YomitanRelive2025
Record Dates: First submitted 2025-09-16; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Metabolic Syndrome; Stress, Psychological
Keywords: Stress reduction; Behavior change; Functional clothing; Exercise; Sleep quality; Heart rate variability; Okinawa; Yomitan
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Stress, Psychological; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups: health information, functional clothing, or moderate exercise.
Masking Description: Due to the nature of the interventions, participants and investigators cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Information Group (Active Comparator): Participants will receive an educational leaflet on lifestyle modification.
  Interventions: Behavioral: Educational Leaflet
- Functional Clothing Group (Experimental): Participants will receive a functional shirt (Relive brand) and will be asked to wear it daily during the 8-week intervention.
  Interventions: Device: Functional Shirt (Relive brand)
- Moderate Exercise Group (Experimental): Participants will receive a structured exercise manual and will be instructed to perform moderate-intensity exercise for 30 minutes, three times per week, for 8 weeks.
  Interventions: Behavioral: Exercise Manual

INTERVENTIONS:
Behavioral: Educational Leaflet — Participants will receive an educational leaflet on lifestyle modification, which provides practical advice on diet, physical activity, and stress management. The leaflet will be distributed at baseline.
  Arms: Health Information Group
Device: Functional Shirt (Relive brand) — Participants will receive a functional shirt designed to support posture and physical comfort (Relive brand). They will be instructed to wear the shirt daily during the 8-week intervention period. Manufacturer: Relive Inc., Japan.
  Arms: Functional Clothing Group
Behavioral: Exercise Manual — Participants will receive a structured exercise manual and will be instructed to perform moderate-intensity exercise (e.g., brisk walking, light jogging, or calisthenics) for 30 minutes, three times per week, over 8 weeks. Weekly follow-up calls or messages will be provided to encourage adherence.
  Arms: Moderate Exercise Group

SUMMARY:
This study is a pilot randomized trial conducted in Yomitan Village, Okinawa, Japan. The purpose is to evaluate whether three simple, low-cost interventions can help reduce stress and support healthy behavior change in community-dwelling adults. The interventions are: (1) providing health information through educational leaflets, (2) wearing functional clothing designed to support physical comfort, and (3) practicing moderate exercise using a simple manual.

A total of 45 adults, aged 20 to 65 years, with overweight or pre-metabolic syndrome will be recruited. Participants will be assigned randomly into one of the three groups. The study duration is eight weeks. Outcomes include fatigue scores, mood states, sleep quality, and heart rate variability measured by a smart ring. Data will be collected at baseline and after eight weeks of intervention.

This study aims to test whether these approaches are feasible, safe, and acceptable for residents. The results will help design larger studies in the future and provide evidence for community-based prevention programs that are easy to adopt in daily life.

DETAILED DESCRIPTION:
Lifestyle-related diseases, including obesity and metabolic syndrome, are major health concerns worldwide. Stress and insufficient physical activity are important risk factors. Developing simple and sustainable interventions that can be adopted in daily life is essential for effective prevention. This feasibility trial compares functional clothing, moderate exercise, and health information in a community setting. The results will provide insight into feasibility, adherence, and potential effectiveness, forming the basis for future large-scale randomized controlled trials and community health programs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 65 years, residing in Yomitan Village
* Body Mass Index (BMI) ≥25, or judged as pre-metabolic syndrome by a physician
* Owns a smartphone and able to use the study application

Exclusion Criteria:

* Severe cardiovascular disease or psychiatric illness
* Medical contraindication to moderate exercise
* Unable to provide informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-04 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Fatigue Score (Visual Analog Scale, 0-100 mm) | Baseline and Week 8
  Change in subjective fatigue measured using a 100-mm Visual Analog Scale (VAS). Scores range from 0 (no fatigue) to 100 (worst possible fatigue). Higher scores indicate worse fatigue.
Total Mood Disturbance (Profile of Mood States-2) | Baseline and Week 8
  Change in total mood disturbance score assessed using the Profile of Mood States-2 (POMS-2). Scores range from -32 to 200. Higher scores indicate worse mood.

SECONDARY OUTCOMES:
Sleep Duration (hours/night) | Baseline and Week 8
  Average nightly sleep duration measured objectively using a smart ring.
Sleep Efficiency (%) | Baseline and Week 8
  Percentage of time in bed spent asleep, measured objectively using a smart ring.
Heart Rate Variability (HRV) | Baseline and Week 8
  Autonomic function assessed via smart ring-derived HRV indicators, including SDNN and RMSSD.
Adherence Rate | Throughout 8-week intervention
  Percentage of participants completing prescribed intervention activities (leaflet reading, shirt wearing, or exercise sessions).
Adverse Events | Throughout 8-week intervention
  Frequency and type of adverse events, including skin irritation and muscle soreness, monitored continuously.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryusei Hospital, Naha, Okinawa, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunton GF, Crosley-Lyons R, Rhodes RE. Affective Response During Real-World Physical Activity as an Intervention Mediator. Exerc Sport Sci Rev. 2023 Oct 1;51(4):140-149. doi: 10.1249/JES.0000000000000321. Epub 2023 May 17. PMID 37195062
- [Background] Stevens CJ, Baldwin AS, Bryan AD, Conner M, Rhodes RE, Williams DM. Affective Determinants of Physical Activity: A Conceptual Framework and Narrative Review. Front Psychol. 2020 Dec 1;11:568331. doi: 10.3389/fpsyg.2020.568331. eCollection 2020. PMID 33335497
- [Background] Dimsdale JE. Psychological stress and cardiovascular disease. J Am Coll Cardiol. 2008 Apr 1;51(13):1237-46. doi: 10.1016/j.jacc.2007.12.024. PMID 18371552
- [Background] Chouchou F, Desseilles M. Heart rate variability: a tool to explore the sleeping brain? Front Neurosci. 2014 Dec 11;8:402. doi: 10.3389/fnins.2014.00402. eCollection 2014. PMID 25565936
- [Background] Cohen S, Janicki-Deverts D, Miller GE. Psychological stress and disease. JAMA. 2007 Oct 10;298(14):1685-7. doi: 10.1001/jama.298.14.1685. No abstract available. PMID 17925521
- See also: Institute for Health Tourism, Ryusei Hospital (project overview) — https://www.ryusei.or.jp/checkup/Consulting#description-con-1